CLINICAL TRIAL: NCT01070277
Title: Antiparasitic Treatment for Returning Travelers With Chronic Diarrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Eli Schwartz MD, DTMH, Director, The Center of Geographic Medicine, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-08-5059-ES-CTIL
Record Dates: First submitted 2010-02-15; First posted 2010-02-18 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Diarrhea; Abdominal Pain; Bloating
Keywords: chronic diarrhea; travelers; Parasites; albendazole; tinidazole
MeSH Terms: conditions — Abdominal Pain | interventions — Tinidazole; Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo arm (Placebo Comparator): 2 placebo pills X2 /day for 2 days followed by
  1 placebo Pill X2 / day for 7 days
  Interventions: Drug: Placebo control
- Tinidazole and Albendazole treatment (Experimental): Tinidazole 1 gram BID for 2 days followed by Albendazole 400mg BID for 7 days
  Interventions: Drug: Tinidazole and Albendazole

INTERVENTIONS:
Drug: Tinidazole and Albendazole — Tinidazole 2 gr/daily for 2 days followed by Albendazole 400mg X2 /day for 7 days
  Arms: Tinidazole and Albendazole treatment
Drug: Placebo control — 2 placebo pills X2 /day for 2 days followed by
  1 placebo Pill X2 / day for 7 days
  Arms: Placebo arm

SUMMARY:
Study hypotheses is that Antiparasitic therapy in patients with chronic diarrhea after travel to a developing country, with a negative stool findings, will be significantly effective in eliminating diarrhea and other gastro-intestinal complaints compared to similar patients receiving placebo.

DETAILED DESCRIPTION:
It is common to encounter travelers from developing countries who suffer from persistent diarrhea after returning home. In many cases repeated stool samples are negative for bacteria, parasites and helminthes and the cause of the diarrhea is not found.

The main debate is whether this condition is a persistent parasitic infection (unidentified) or post-infectious irritable bowel syndrome.However, clinical experience suggests that some of these travelers respond to antiparasitic therapy.

This study aims to answer the question whether antiparasitic treatment in these cases is beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Diarrhea (3 or more soft stools per day) for at least two weeks after a trip to a developing country in the past year
* Stool sample negative for bacteria, parasites and helminthes at least once
* Has not received, until now, antiparasitic or antihelminthic therapy

Exclusion Criteria:

* Bloody diarrhea
* Fever during enrolment 5. Allergy to the offered medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
improvement in gastrointestinal complaints | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Chaim Sheba Medical Center, Tel Hashomer, Israel, Ramat Gan
  - Sheba Medical Center, Ramat Gan